CLINICAL TRIAL: NCT03345589
Title: A Randomized Controlled Trial of 18-22mg/kg/d Ursodeoxycholic in Refractory Primary Biliary Cholangitis
Brief Title: A Trial of 18-22mg/kg/d Ursodeoxycholic in Refractory Primary Biliary Cholangitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Li Yang, Principal Investigator, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC-3
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Primary Biliary Cholangitis
Keywords: Ursodeoxycholic Acid
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 18-22mg/kg/d Ursodeoxycholic group (Experimental)
  Interventions: Drug: 18-22mg/kg/d Ursodeoxycholic
- 13-15mg/kg/d Ursodeoxycholic group (Placebo Comparator)
  Interventions: Drug: 13-15mg/kg/d Ursodeoxycholic

INTERVENTIONS:
Drug: 18-22mg/kg/d Ursodeoxycholic — 18-22mg/kg/d Ursodeoxycholic
  Arms: 18-22mg/kg/d Ursodeoxycholic group
Drug: 13-15mg/kg/d Ursodeoxycholic — 13-15mg/kg/d Ursodeoxycholic
  Arms: 13-15mg/kg/d Ursodeoxycholic group

SUMMARY:
This study evaluates the effect of 18-22mg/kg/d Ursodeoxycholic in refractory Primary Biliary Cholangitis

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary biliary cholangitis
* Treated with Ursodeoxycholic Acid in West China Hospital for at least 6 month and suboptimal response to Ursodeoxycholic Acid

Exclusion Criteria:

* Autoimmune hepatitis
* Primary sclerosing cholangitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Percent of patients that achieve biochemical remission of primary biliary cholangitis(PBC) | Month 6 during treatment with 13-15mg/kg/d ursodeoxycholic acid or 18-22mg/kg/d ursodeoxycholic acid
  Percent of patients that achieve biochemical remission of primary biliary cholangitis(PBC) in two arms.

SECONDARY OUTCOMES:
Alkaline phosphatase | Week 2 and Month 1, 3, 6,9,12
  (ALP)
Glutamyltransferase | Week 2 and Month 1, 3, 6,9,12
  (GGT)
Alanine transaminase | Week 2 and Month 1, 3, 6
  (ALT)
Aspartate transaminase | Week 2 and Month 1, 3, 6, 9,12
  (AST)
Total bilirubin | Week 2 and Month 1, 3, 6, 9,12
  (TB)

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, MD, Study Chair — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China